CLINICAL TRIAL: NCT03265873
Title: Contribution of the ENT Surgeon's Clinical Evaluation to the Contouring of Target Volumes and Organs Eligible for Radiotherapy in Head and Neck Cancers
Brief Title: Contribution of the ENT (Ear, Nose, and Throat) Surgeon's Clinical Evaluation to the Contouring of Target Volumes and Organs Eligible for Radiotherapy in Head and Neck Cancers
Acronym: CONTOUR
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: DBU_2017_13
Record Dates: First submitted 2017-08-28; First posted 2017-08-29 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Radiotherapy, Conformal (IMRT); Head and Neck Cancer; Otolaryngology; Surgeons; Radiation Oncologists
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Systematic consideration of the advice of the ENT surgeon in the determination of the radiotherapy target volumes in head and neck cancers. — The contouring of the different target volumes will be first performed by the radiotherapists. During the Head and Neck Tumor Board, the volumes initially determined by the radiotherapists will be analyzed jointly by the radiotherapists and the patient's ENT surgeon to carry out, if necessary, modifications, taking into account clinical observations, intraoperative findings (if any) and endoscopy findings. Concordance parameters will be calculated in a second time with the determined volumes (in particular, index of concordance, coefficient of similarity).

SUMMARY:
Radiotherapy (RT), surgery and chemotherapy (CT) are treatments for head and neck cancers, used alone or in combination. Conformal RT with Intensity Modulation (IMRT) is currently the reference technique. IMRT requires a precise definition of the target volumes to be treated and the anatomical structures to be protected from irradiation. Most studies of head and neck cancers published in the literature demonstrate the variability in the contouring of the target volumes between radiotherapists. This may have an impact on dosimetry. To date, no studies have evaluated the impact of the ENT surgeon's evaluation in volumes contouring. The aim of this study is to compare the volumes determined by the radiotherapists alone and those determined jointly by the radiotherapists and the ENT surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Cancer of the upper aerodigestive tract (oral cavity, oropharynx, larynx, hypopharynx, rhinopharynx, salivary glands, facial sinuses, orbital cavity, ear);
* Cancer confirmed by histopathological analysis;
* Therapeutic protocol including radiotherapy.

Exclusion Criteria:

* Any history of radiotherapy of the head and neck
* Synchronous head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with head and neck cancer who require radiotherapy.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with head and neck cancer for whom a change in the CTV (Clinical Target Volume) was made following the advice of the ENT surgeon. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Clément, MD, Principal Investigator — Hôpital d'Instruction des armées Percy
Locations (2):
- France (2):
  - Hôpital d'Instruction des Armées, Clamart
  - Fondation Ophtalmologique A. de Rothschild, Paris

IPD SHARING:
Plan to Share IPD: Undecided